CLINICAL TRIAL: NCT05090436
Title: Schroth Exercise Versus Functional Electrical Stimulation in Adolescent With Spinal Deformities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Delta University for Science and Technology (Other)
Responsible Party: Principal Investigator, Amira Hussin Hussin Mohammed, Assistant. Professor of physical therapy, Department of Physical Therapy for Pediatrics, Delta University for Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: schroth exercises
Record Dates: First submitted 2021-09-17; First posted 2021-10-22 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Idiopathic Spinal Deformities
MeSH Terms: interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Schroth Exercise (Experimental): The Schroth Method is a nonsurgical option for scoliosis treatment. It uses exercises customized for each patient to return the curved spine to a more natural position. The goal of Schroth exercises is to de-rotate, elongate and stabilize the spine in a three-dimensional plane. it will be applied 3 session per week for 3 months.
  Interventions: Other: Schroth Exercise
- Functional Electrical Stimulation (Experimental): 30 minutes of Functional Electrical Stimulation (FES) three times a week for 3 months. Two electrodes were attached on the lateral parts of the convex side of the body, and two others on the erector spinae muscles. FES (CU-FS1; Novastim, Korea) was set at a frequency of 35 Hz, with a 250-μs pulse width. Electrical stimulation lasted for 6 seconds, followed by a 6-second rest.
  Interventions: Other: Functional Electrical Stimulation (physiotherapy techniques)

INTERVENTIONS:
Other: Schroth Exercise — two month (three session per week)
  Arms: Schroth Exercise
Other: Functional Electrical Stimulation (physiotherapy techniques) — two month (three session per week)
  Arms: Functional Electrical Stimulation

SUMMARY:
Abnormal spinal curvature can occur as a result of neurologic, orthopedic or idiopathic factors. The role of physiotherapy is not only to prevent intrinsic changes that may occur in the spine but also be used to correct postural abnormalities. this study will investigate the impact of Schroth Exercise compared to Functional Electrical Stimulation in Adolescent With Spinal Deformities (scoliosis and or kyphosis).

ELIGIBILITY:
Inclusion Criteria:

* Children in this group will be healthy category according to CDC (Centers for Disease Control and Prevention) growth chart which ranged from BMI-for-age 5th to 85th percentiles .
* All children are normal &perform all activities of daily living
* They were able to understand and follow verbal commands and instructions included in the testing procedures.

Exclusion Criteria:

* All of them could be part of recreational activities in their public schools but no competitive sports.
* Children who participated in any regular sport activities involving the lower extremities will be excluded.
* None of them had any surgical intervention .
* None of them had any history of other musculoskeletal deformities or neuromuscular disorders.
* They had neither visual, auditory defect.

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2021-10-25 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
cobb angle | at the beginning of the study
  The measurement of Cobb angle involves estimating the angle between the two tangents of the upper and lower end-plates of the upper and lower end vertebra, respectively.
cobb angle | by the end of successful two month of intervention
  The measurement of Cobb angle involves estimating the angle between the two tangents of the upper and lower end-plates of the upper and lower end vertebra, respectively

CONTACTS AND LOCATIONS:
Locations (1):
- Amira Hussin Mohammed, Gamasa, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR